CLINICAL TRIAL: NCT01576250
Title: The Effect of Lowered Physical Activity (Induced by Lower Limb Suspension (ULLS)) on Insulin Sensitivity and Lipid and Glucose Metabolism
Brief Title: The Effect of Lowered Physical Activity on Insulin Sensitivity and Lipid and Glucose Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Principal Investigator, Lena Bilet, PhD student, Maastricht University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: NL38795.068.11/METC 11-3-074
Record Dates: First submitted 2012-04-10; First posted 2012-04-12 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Insulin Sensitivity
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- unilateral lower limb suspension (Experimental): This is an intervention study, where each subject will undergo 12 days of unilateral lower limb suspension. Randomly, the dominant or the non-dominant leg of the subject will be suspended by attachment of a sling to a non-rigid ankle brace and to a harness on the upper body and unloaded from all weight bearing. The knee will be slightly flexed at an angle of 130°. Hip, knee and ankle will be fully mobile. The sling will be used during all locomotory activity, and the subjects will use crutches for walking.
  Interventions: Other: unilateral lower limb suspension

INTERVENTIONS:
Other: unilateral lower limb suspension — This is an intervention study, where each subject will undergo 12 days of unilateral lower limb suspension. Randomly, the dominant or the non-dominant leg of the subject will be suspended by attachment of a sling to a non-rigid ankle brace and to a harness on the upper body and unloaded from all weight bearing. The knee will be slightly flexed at an angle of 130°. Hip, knee and ankle will be fully mobile. The sling will be used during all locomotory activity, and the subjects will use crutches for walking.

SUMMARY:
The purpose of this study is to investigate the effects of lowered physical activity (resulting in decreased muscle mitochondrial oxidative capacity) alone and together with increased plasma free fatty acid availability (by infusion of a clinically widely used lipid emulsion (Intralipid)) on insulin sensitivity and glucose and lipid metabolism. To this end, we will compare skeletal muscle insulin sensitivity and glucose and lipid metabolism (within one subject) after 9 days of immobilization of one leg (unilateral lower limb suspension(ULLS))(decreased muscle mitochondrial oxidative capacity) versus an active control leg (unchanged muscle mitochondrial oxidative capacity). Further, changes in IMCL and fatty acid intermediates will be investigated in the immobilized vs the control leg, and this will be related to insulin sensitivity. The effectiveness of the ULLS intervention will be tested by measuring muscle mitochondrial oxidative capacity in both the immobilized and the control leg. All measurements will be performed both in the immobilized and control leg after 9 days of ULLS.

DETAILED DESCRIPTION:
In the Netherlands and worldwide, the number of individuals suffering from obesity and type 2 diabetes mellitus is rising steadily. It is well established that obesity predisposes individuals to accumulation of excessive fat in non-adipose tissues such as the liver, the heart and skeletal muscle (called steatosis or ectopic fat accumulation). Furthermore, in sedentary humans ectopic fat accumulation in skeletal muscle is strongly associated with insulin resistance. However, paradoxically, IntraMyoCellular Lipid (IMCL) content is also increased in highly insulin sensitive endurance trained subjects (known as the athlete's paradox). This is suggesting that IMCL per se is not causative in skeletal muscle insulin resistance. The increased IMCL storage following endurance training serves to match training-induced increase in oxidative capacity and reliance on fat as a substrate during exercise, whereas in obesogenic/diabetogenic conditions the high fat availability is not matched by improved oxidative capacity. It is therefore speculated that under the latter conditions, the lipid intermediates of IMCL metabolism such as diacylglycerol (DAG), ceramides and fatty acyl-CoAs will accumulate and impede cellular insulin signalling. The rate of oxidative capacity is regulated by mitochondria, which are cellular organelles responsible for cellular energy production and cellular metabolism. Therefore, the overall hypothesis of this project is that a low muscle mitochondrial oxidative capacity can lead to muscle fat accumulation and/or accumulation of lipid intermediates when fatty acid availability is high, and this may result in insulin resistance in skeletal muscle.

ELIGIBILITY:
Inclusion Criteria:

* Men between 18-35 years of age at time of enrolment
* Non smoking
* No recent bone fractures of the limbs
* No cardiovascular medication or other medication
* No family history of thrombosis
* No engagement in programmed exercise for more than two hours a week
* Stable dietary habits
* No contra-indication for MRI

Exclusion Criteria:

* Regular smokers
* Participation in other studies
* Female sex
* Recent bone fractures of the limbs
* Medication use
* Cardiovascular disease
* Family history of type 2 diabetes mellitus
* Family history of thrombosis
* Contraindications for MRS scans:
* Electronic implants such as pacemakers or neurostimulator
* Iron-containing foreign bodies in eyes or brain
* Some hearing aids and artificial (heart) valves which are contraindicated for MRS
* Claustrophobia
* Participants, who do not want to be informed about unexpected medical findings, or do not wish that their physician will be informed, cannot participate in the study

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2012-04; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity | after 9 days of ULLS
  After 9 days of ULLS a muscle biopsy will be derived before and after a 5 h lipid infusion,from both the immobilized and the control leg. Insulin sensitivity will further be investigated from the skeletal muscle tissue ex vivo.

SECONDARY OUTCOMES:
intramyocellularlipid content | after 9 days of ULLS
  After 9 days of ULLS a muscle biopsy will be derived before and after a 5 h lipid infusion,from both the immobilized and the control leg. Muscle tissue will immediately be frozen and stored for later determination of Intramyocellular lipid content.
Lipid intermediates | after 9 days of ULLS
  After 9 days of ULLS a muscle biopsy will be derived before and after a 5 h lipid infusion,from both the immobilized and the control leg. Lipid intermediates will further be investigated from the skeletal muscle tissue ex vivo.
Lipid metabolism | after 9 days of ULLS
  After 9 days of ULLS a muscle biopsy will be derived before and after a 5 h lipid infusion,from both the immobilized and the control leg. Lipid metabolism will further be investigated from the skeletal muscle tissue ex vivo.
Glucose metabolism | after 9 days of ULLS
  After 9 days of ULLS a muscle biopsy will be derived before and after a 5 h lipid infusion,from both the immobilized and the control leg. Glucose metabolism will further be investigated from the skeletal muscle tissue ex vivo.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Schrauwen, Ph.D., Study Director — Maastricht University Medical Center (MUMC); Lena Bilet, MSc., Principal Investigator — Maastricht University Medical Center (MUMC)
Locations (1):
- Maastricht University Medical Center, Maastricht, Netherlands

REFERENCES:
- [Derived] Bilet L, Phielix E, van de Weijer T, Gemmink A, Bosma M, Moonen-Kornips E, Jorgensen JA, Schaart G, Zhang D, Meijer K, Hopman M, Hesselink MKC, Ouwens DM, Shulman GI, Schrauwen-Hinderling VB, Schrauwen P. One-leg inactivity induces a reduction in mitochondrial oxidative capacity, intramyocellular lipid accumulation and reduced insulin signalling upon lipid infusion: a human study with unilateral limb suspension. Diabetologia. 2020 Jun;63(6):1211-1222. doi: 10.1007/s00125-020-05128-1. Epub 2020 Mar 17. PMID 32185462